CLINICAL TRIAL: NCT03088202
Title: PALLiON - PALLiative Care In ONcology - a Cluster-randomized Trial to Improve the Care for Cancer Patients With a Short Life Expectancy
Brief Title: PALLiON - PALLiative Care In ONcology
Acronym: PALLiON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Principal Investigator, Marianne Jensen Hjermstad, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016/1220REK
Record Dates: First submitted 2017-01-30; First posted 2017-03-23 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Neoplasia Prostate
Keywords: cancer; palliative care; PROMs; survival; QoL; referral
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Masking Description: No masking, the randomization applies to institutions, not patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Educational program Standardized care pathways Early palliative care
  Interventions: Other: Educational program; Other: Standardized care pathways; Other: Early palliative care
- Control arm (No Intervention): Usual care

INTERVENTIONS:
Other: Educational program — E-learning lectures, group exercises, skills training
  Arms: Intervention arm
Other: Standardized care pathways — Pathways for systematic follow-up
  Arms: Intervention arm
Other: Early palliative care — Compulsory referral to palliative care at inclusion
  Arms: Intervention arm

SUMMARY:
A major concern in today's oncology is the complexity of treatment that increases costs. A main contributor is the increasing use of chemo- and radiotherapy during end of life (EoL: the last 12 months of life). Importantly, intensive chemotherapy in EoL has uncertain efficacy, may result in frequent hospitalizations and less time spent at home. Also, patients with incurable disease who receive intensive treatment at EoL have worse quality of life (QoL). A systematic palliative care (PC) approach that focuses on optimal symptom management and maintenance of QoL of patients and family is often introduced too late in the disease trajectory. Studies indicate that early introduction of PC in patients with unfavorable prognosis may improve QoL and other symptoms and prolong survival. These and related findings have made international stakeholders advocate a stronger integration of oncology and PC for patients with incurable cancer.

The present project is a national multicenter cluster-randomized trial (RCT) in 12 oncology departments in all 4 Norwegian health regions. The project tests the efficacy of a complex tripod intervention that integrates oncology and PC for cancer patients with a life-expectancy <12 months who receive chemotherapy and includes: A) systematic electronic assessment of symptoms, B) implementation of standardized care pathways and C) an education program for oncologists/PC physicians. The PC pathway focuses on the patient's journey through the PC trajectory including EoL care in order to improve quality of care and reduce the variability in clinical practice and costs. The intervention aims at empowering physicians, patients and relatives and promoting shared-decision-making.

DETAILED DESCRIPTION:
Patients with incurable disease who receive intensive treatment at EoL have worse quality of life (QoL) compared with those receiving symptomatic treatment. Also, a PC approach at an early stage in patients with unfavorable prognosis may improve patients' QoL and symptom control, may lead to prolonged survival and give patients and caregivers a more realistic perspective on the disease and prognosis. Further, there is documentation that caregivers of patients with advanced cancer are generally more satisfied and report less depressive symptoms with an early introduction of PC.

These and related findings in the wake of a study (NEJM 2010) initiated the current debate and have made international stakeholders advocate a stronger integration of oncology and PC for patients with incurable cancer. Despite a rapid development of PC services during the last 15-20 years, there is still a distinct separation between oncology and PC in Norway as in other Western countries. This infers that the potential for optimal care during the last phase of life for those patients has not been fully explored, despite the documented advantages for both patients and caregivers. However, results from studies on integration of oncology and PC from other countries e.g. the USA, may not be directly transferable to Norway, given the different health care organizations, reimbursement issues and the different indications for and the high degree of hospice use.

Information given to cancer patients and caregivers about the disease and its treatment is important at all stages of disease, and is crucial in relation to PC in order to facilitate shared decision making, and improve satisfaction with care, patients' sense of control, QoL and communication with patient and caregivers. As PC also aims to improve the QoL of caregivers waiting to include caregivers until patients are in their last weeks or days of life may not adequately address patient or caregiver distress. Further, the benefits of early integration of PC on caregiver's distress and QoL remain inconclusive.

Thus, the overall aim of PALLiON is to improve the quality and efficacy of cancer care by implementing an early integration of oncology and PC in patients with advanced cancer who receive chemotherapy. The long-term objective is a change of today's oncology practice. Today, the method of referral to PC is most often based on care needs in contrast to referrals based on diagnosis and prognosis used in the RCTs that have documented favorable results. As we know that the timing of referral is important to optimize the benefits of PC, we aim to change this practice.

The implementation method in PALLiON is a complex intervention consisting of a) a structured educational program for oncologists, palliative care physicians and nurses, b) standardized care pathways with a systematic integration of oncology and palliative care for each of the included cancer diagnoses, and c) systematic use of Eir - an electronic assessment tool for patient-reported outcomes (PROMs), in the standardized care pathways, combined with evidence-based treatment recommendations in the clinical consultations.

The design makes it possible to evaluate the effect of an early integration of oncology and PC at the institutional and patient levels between the intervention and control arms. Further, a potential effect of the intervention at each of the centers in the intervention arm can be evaluated by comparing the post-intervention data with historical data e.g. on use of chemotherapy, number of re-admissions / emergency admissions in the very last stages of life as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* A verified metastatic or locally advanced cancer of the upper GI tract, lower GI tract, pancreas, liver, breast, bladder, prostate, kidney, cholangiocarcinoma, or malignant melanoma
* Defined as a palliative care patient, with expected life expectancy of <12 months
* Scheduled to start what is perceived as last line of chemotherapy (definition: tumor directed medical therapy)

  o Observe: different time points for inclusion and line of treatment apply for the specific diagnoses
* Age > 18 years
* Fluency in written and oral Norwegian
* Physically and cognitively able to provide written informed consent, based on clinical judgment
* Scheduled to receive all oncological and specialized palliative treatment at the participating hospital
* World Health Organization (WHO) performance status 0-2

Exclusion Criteria:

* Any serious psychiatric diagnosis (e.g. psychotic, bipolar disorder), substance abuse or cognitive impairment as judged by standard clinical criteria (disturbed consciousness, disorientation to time/place and attention deficits) at the discretion of the attending physician that precludes completion of PROs
* A cancer diagnosis other than the ones above
* Multiple malignancies
* Serious substance abuse
* Already included in a palliative care program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 659 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Use of chemotherapy | 3 months before death
  Number of patients who receive chemotherapy during their last 3 months of life

SECONDARY OUTCOMES:
Initiation and discontinuation of chemotherapy | 3 months before death
  Number of patients who start and discontinue chemo, and number of cycles
Use of artificial nutrition | 1 month before death
  Number of patients who receive artificial nutrition during their last month of life
Use of concomitant medication | 1 month before death
  Number of patients who receive concomitant medication during their last month of life

CONTACTS AND LOCATIONS:
Overall Officials: Jon H Loge, PhD, Principal Investigator — Professor
Locations (12):
- Norway (12):
  - University Hospital of North Norway, Tromsø, Troms
  - Ålesund Hospital Trust, Ålesund
  - Nordland Hospital Trust, Bodø
  - Østfold Hospital Trust, Fredrikstad
  - Førde Hospital Trust, Førde
  - Sørlandet Hospital Trust, Kristiansand
  - Akershus University Hospital, Oslo
  - Oslo University Hospital, Oslo
  - Telemark Hospital Trust, Skien
  - Stavanger University Hospital, Stavanger
  - Norwegian University of Science and Technology, Trondheim
  - Vestfold Hospital trust, Tønsberg

IPD SHARING:
Plan to Share IPD: Yes
If desired, other collaborators may use data collected at their own institution. However, this is subject to approval from the study scientific committee, and only applies after publication of the main study publication
Supporting Information: Study Protocol, SAP
Time Frame: end 2019
Access Criteria: co-authorship use of own data for quality assurance / publications

REFERENCES:
- [Derived] Hjermstad MJ, Pirnat A, Aass N, Andersen S, Astrup GL, Dajani O, Garresori H, Guldhav KV, Hamre H, Haukland EC, Jordal F, Lundeby T, Lohre ET, Mjaland S, Paulsen O, Semb KA, Staff ES, Wester T, Kaasa S. PALLiative care in ONcology (PALLiON): A cluster-randomised trial investigating the effect of palliative care on the use of anticancer treatment at the end of life. Palliat Med. 2024 Feb;38(2):229-239. doi: 10.1177/02692163231222391. Epub 2024 Jan 9. PMID 38193250
- [Derived] Lundeby T, Finset A, Kaasa S, Wester TE, Hjermstad MJ, Dajani O, Wist E, Aass N. A complex communication skills training program for physicians providing advanced cancer care - content development and barriers and solutions for implementation. J Commun Healthc. 2023 Mar;16(1):46-57. doi: 10.1080/17538068.2022.2039468. Epub 2022 Feb 20. PMID 36919800
- [Derived] Hjermstad MJ, Aass N, Andersen S, Brunelli C, Dajani O, Garresori H, Hamre H, Haukland EC, Holmberg M, Jordal F, Krogstad H, Lundeby T, Lohre ET, Mjaland S, Nordbo A, Paulsen O, Schistad Staff E, Wester T, Kaasa S, Loge JH. PALLiON - PALLiative care Integrated in ONcology: study protocol for a Norwegian national cluster-randomized control trial with a complex intervention of early integration of palliative care. Trials. 2020 Apr 2;21(1):303. doi: 10.1186/s13063-020-4224-4. PMID 32241299